CLINICAL TRIAL: NCT04089475
Title: Hypo-pigmented Skin Lesions in Children : Dermoscopic Evaluation
Brief Title: Dermoscopy of Hypo-pigmented Lesions in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, SNIsrael, principal investigator, Assiut University
Other Study IDs: DHLC
Record Dates: First submitted 2019-09-11; First posted 2019-09-13 (Actual); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Hypopigmented Skin
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Dermoscope — Dermoscopy is a noninvasive diagnostic tool that permits the visualization of morphological features that are not visible to the naked eye thus representing a link between macroscopic clinical dermatology and microscopic dermatopathology.

SUMMARY:
Hypo-pigmented skin lesions in children are of great concern in the society. They cause anxiety among children and their parents due to the social stigma attached to these conditions especially in dark skinned children. Hypo pigmented skin lesions are commonly encountered in day-to-day practice, and they pose a diagnostic challenge for the clinician. They are one of the commonest complains in the dermatology clinics and generally share the same patient complaint which is characterized by the presence of hypo or depigmented patches or macules .

Dermoscopy may be a helpful as a non-invasive tool in assisting the differential diagnosis of several hypopigmented macular lesions and has the potential to improve the diagnostic accuracy.

DETAILED DESCRIPTION:
Among the most common disorders of hypo-pigmentation in children are pityriasis alba, vitiligo, nevus depigmentosus, postinflammatory hypopigmentation and tinea versicolor ; while idiopathic guttate hypomelanosis and hypopigmented mycosis fungoides comes late.

Pityriasis alba : is a low-grade type of eczema/dermatitis mostly occurring in children and young adults , usually seen as dry, fine-scaled, pale patches on the face .

Vitiligo : is an acquired, autoimmune, idiopathic disorder characterized by circumscribed depigmented macules and patches with or without leukotrichia .

Nevus depigmentosus : is a localized hypopigmentation which most of the time is congenital. It is considered as a form of cutaneous mosaicism.

Postinflammatory hypopigmentation : is an acquired partial or total loss of skin pigmentation occurring after cutaneous inflammation. Many cutaneous inflammatory conditions lead to postinflammatory hypopigmentation in children as :Atopic dermatitis , Insect bite reactions, Psoriasis, Stevens-Johnson syndrome ….; Infections as Chickenpox, Impetigo …..; Cutaneous injuries from burns, irritants .All tend to induce postinflammatory hypopigmentation rather than hyperpigmentation .

Pityriasis versicolor or tinea versicolor : is a fungal infection of the superficial layer of skin caused by Malassezia yeasts. It is clinically characterized by hyperpigmented or hypopigmented, round to oval lesions covered with scales commonly found on the trunk, upper arms and face. Although it's common in adults but it can be seen in older group of children .

Idiopathic guttate hypomelanosis : is an acquired leukoderma found in all races; Its pathogenesis is unknown but may depend on various factors such as patient age and sun-exposure. Clinically, the lesions are porcelain-white macules, usually 2-6 mm in size, but sometimes they are larger. The borders are sharply defined, often angular and irregular with normal skin markings.

Mycosis fungoides, the most common primary cutaneous T-cell lymphoma: is a neoplastic disease characterized by classical non-infiltrated lesions (patches), plaques, tumors, and erythrodermic stages .It is considered a serious condition that has been seen before in children. Hypopigmented mycosis fungoides is one of its variants that is presented by hypopigmented-to-achromic lesions, sometimes with a vitiligo-like aspect.

In addition to clinical picture, Woods light examination and potassium hydroxide scrapping for scaly hypopigmented macules and histopathological evaluation are used to be the gold standard tests for diagnosis of those hypopigmented lesions in children.

Dermoscopy is a noninvasive diagnostic tool that permits the visualization of morphological features that are not visible to the naked eye thus representing a link between macroscopic clinical dermatology and microscopic dermatopathology . Recently, awareness and knowledge of dermoscopy have increased tremendously in many countries in diagnosis of many skin conditions .

Dermoscopy may be a helpful as a non-invasive tool in assisting the differential diagnosis of several hypopigmented macular lesions and has the potential to improve the diagnostic accuracy. New studies have documented dermoscopic features in vitiligo , While very few reports have documented the dermoscopic features of the other hypopigmented lesions.

ELIGIBILITY:
Inclusion Criteria:

* All children up to (18) years old attending Assiut University Hospital complaining of hypopigmented skin lesions.

Exclusion Criteria:

* Patients on topical or systemic treatment ( in the last 1 and 3 months , respectively) will be excluded.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children up to (18) years old attending Assiut University Hospital complaining of hypopigmented skin lesions.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
To detect the sensitivity and specificity of the dermoscope in diagnosis of hypopigmented skin lesions in children | Almost 6 months after we start
  correlate the diagnosis of the hypopigmented lesions with the dermoscopic features and test the validity of the dermoscope in diagnosis .

REFERENCES:
- [Background] Das JK, Gangopadhyay AK. Mycosis fungoides with unusual vitiligo-like presentation. Indian J Dermatol Venereol Leprol. 2004 Sep-Oct;70(5):304-6. PMID 17642645
- [Background] Al-Refu K. Dermoscopy is a new diagnostic tool in diagnosis of common hypopigmented macular disease: A descriptive study. Dermatol Reports. 2018 Dec 21;11(1):7916. doi: 10.4081/dr.2018.7916. eCollection 2019 Jan 23. PMID 31119026
- [Background] Kim SK, Kang HY, Lee ES, Kim YC. Clinical and histopathologic characteristics of nevus depigmentosus. J Am Acad Dermatol. 2006 Sep;55(3):423-8. doi: 10.1016/j.jaad.2006.04.053. Epub 2006 May 30. PMID 16908347
- [Background] Kim SK, Kim EH, Kang HY, Lee ES, Sohn S, Kim YC. Comprehensive understanding of idiopathic guttate hypomelanosis: clinical and histopathological correlation. Int J Dermatol. 2010 Feb;49(2):162-6. doi: 10.1111/j.1365-4632.2009.04209.x. PMID 20465639
- [Background] Lallas A, Giacomel J, Argenziano G, Garcia-Garcia B, Gonzalez-Fernandez D, Zalaudek I, Vazquez-Lopez F. Dermoscopy in general dermatology: practical tips for the clinician. Br J Dermatol. 2014 Mar;170(3):514-26. doi: 10.1111/bjd.12685. PMID 24266695
- [Background] Miazek N, Michalek I, Pawlowska-Kisiel M, Olszewska M, Rudnicka L. Pityriasis Alba--Common Disease, Enigmatic Entity: Up-to-Date Review of the Literature. Pediatr Dermatol. 2015 Nov-Dec;32(6):786-91. doi: 10.1111/pde.12683. Epub 2015 Oct 19. PMID 26477326
- [Background] Pedrosa AF, Lisboa C, Goncalves Rodrigues A. Malassezia infections: a medical conundrum. J Am Acad Dermatol. 2014 Jul;71(1):170-6. doi: 10.1016/j.jaad.2013.12.022. Epub 2014 Feb 22. PMID 24569116
- [Background] Thatte SS, Khopkar US. The utility of dermoscopy in the diagnosis of evolving lesions of vitiligo. Indian J Dermatol Venereol Leprol. 2014 Nov-Dec;80(6):505-8. doi: 10.4103/0378-6323.144144. PMID 25382506
- [Background] Yamashita T, Abbade LP, Marques ME, Marques SA. Mycosis fungoides and Sezary syndrome: clinical, histopathological and immunohistochemical review and update. An Bras Dermatol. 2012 Nov-Dec;87(6):817-28; quiz 829-30. doi: 10.1590/s0365-05962012000600001. PMID 23197199
- [Background] Vachiramon V, Thadanipon K. Postinflammatory hypopigmentation. Clin Exp Dermatol. 2011 Oct;36(7):708-14. doi: 10.1111/j.1365-2230.2011.04088.x. Epub 2011 Jun 14. PMID 21671990
- [Background] Sori T, Nath AK, Thappa DM, Jaisankar TJ. Hypopigmentary disorders in children in South India. Indian J Dermatol. 2011 Sep-Oct;56(5):546-9. doi: 10.4103/0019-5154.87152. PMID 22121275
- [Background] Argenziano G, Soyer HP, Chimenti S, Talamini R, Corona R, Sera F, Binder M, Cerroni L, De Rosa G, Ferrara G, Hofmann-Wellenhof R, Landthaler M, Menzies SW, Pehamberger H, Piccolo D, Rabinovitz HS, Schiffner R, Staibano S, Stolz W, Bartenjev I, Blum A, Braun R, Cabo H, Carli P, De Giorgi V, Fleming MG, Grichnik JM, Grin CM, Halpern AC, Johr R, Katz B, Kenet RO, Kittler H, Kreusch J, Malvehy J, Mazzocchetti G, Oliviero M, Ozdemir F, Peris K, Perotti R, Perusquia A, Pizzichetta MA, Puig S, Rao B, Rubegni P, Saida T, Scalvenzi M, Seidenari S, Stanganelli I, Tanaka M, Westerhoff K, Wolf IH, Braun-Falco O, Kerl H, Nishikawa T, Wolff K, Kopf AW. Dermoscopy of pigmented skin lesions: results of a consensus meeting via the Internet. J Am Acad Dermatol. 2003 May;48(5):679-93. doi: 10.1067/mjd.2003.281. PMID 12734496